CLINICAL TRIAL: NCT00911469
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre, Single and Multiple Ascending Dose Study of AS902330 (rhFGF-18) Administered Intra-articularly in Patients With Knee Primary Osteoarthritis Who Are Candidates for Total Knee Replacement.
Brief Title: Study of AS902330 (rhFGF-18) Administered Intra-articularly in Patients With Knee Primary Osteoarthritis Who Are Candidates for Total Knee Replacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27575
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; fibroblast growth factor 18
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AS902330
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AS902330 — 3, 10, 30, 100 or 300 µg intra-articular injection per subject in the Single Ascending Dose (SAD) cohorts and 10, 30, 100, 300 µg or highest tolerated dose intra-articular injection per week for three weeks per subject in the Multiple Ascending Dose (MAD) cohorts.
  Arms: 1
Drug: Placebo — Placebo or, 3, 10, 30, 100 or 300 µg intra-articular injection per subject in SAD cohorts and placebo or, 10, 30, 100, 300 µg or highest tolerated dose of AS902330 intra-articular injection per week for three weeks per subject in MAD cohorts.
  Arms: 2

SUMMARY:
Osteoarthritis (OA) is one of the most common diseases affecting the joints, usually those that are weight bearing such as the knees. OA is considered to be a disease of the cartilage in the joints even though it involves the whole joint, including the bone and synovium (thin lining of the joints which produces synovial fluid). With time, more and more of the cartilage is destroyed by the disease with inflammation commonly occurring.

AS902330 is expected to increase the production and development of specific bone cells: chondrocytes and osteoblasts (cells that produce and maintain bone and cartilage). This is expected to lead to repair and regeneration of the cartilage, and a narrowing of the space width between the knee joints in a selected region of the knee.The purpose of this study is to see how safe treatment with AS902330 is, and to evaluate its effect on the knee cartilage. In addition, the study will also measure the effects of AS902330 in the blood.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of knee primary femoro-tibial OA by standard American College of Rheumatology Criteria (ACR) for at least six months (clinical AND radiological criteria)
2. Postmenopausal or surgically sterile female ≥ 40 years of age Post-menopausal status will be confirmed by no menstrual periods for 12 consecutive months and no other biological or physiological cause for amenorrhea can be identified or Male ≥ 40 years of age willing to use contraception (condom with spermicide) from the first day of treatment until 2 months after the end of the treatment (3rd injection in Period 2) Even though systemic exposure of the drug is not foreseen at the doses used in this study, due to the absence of data on teratogenic potential of the drug, a very conservative approach on contraception is taken based on the spermatogenesis duration in humans.
3. Candidate for Total Knee Replacement in the target knee, according to NIH consensus statement on Total Knee Replacement (2003)
4. Date of planned Total Knee Replacement in the target knee ≥ 2 weeks after the anticipated last injection of study drug
5. Subjects may be on treatment for symptomatic relief of OA, including NSAIDs (including Cox2 specific inhibitors); for NSAIDs, the dose should be stable for 4 weeks before baseline and during the study until day 4 after last injection. Paracetamol/acetaminophen (according to local standards and up to 4 grams per day) is allowed as rescue medication
6. Willingness to stay in hospital for 24h after injection for SAD regimens and after first injection for MAD regimens (and up to 4 hours after second and third injections for MAD regimens) for safety and PK evaluation
7. Willingness to complete a diary card to evaluate local tolerability and adverse events throughout the study
8. Subjects must have read and understood the informed consent form and must have signed it prior to any study related procedure
9. Subjects must fully understand the requirements of the study and be willing to comply with all study visits and assessments

Exclusion Criteria:

1. Any condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation
2. Clinically significant abnormal hematology or biochemistry values (platelets, hemoglobin, leucocytes, alkaline phosphatase, AST, ALT, blood creatinine, bilirubin)
3. Receipt of any investigational product or any experimental therapeutic procedure within the last 12 weeks preceding screening
4. Intra-articular treatment with steroids or hyaluronic acid derivatives within the past 3 months (systemic symptomatic treatments with NSAIDs are allowed when stable for 4 weeks prior to first injection)
5. Planned major surgery (e.g. joint replacement) within 2 weeks after last injection
6. History of previous surgery (TKR or partial knee replacement) on the target knee
7. Lesions at the planned injection site that would present a contra-indication to local injection of the study drug (e.g., open wounds and infections of the skin)Any drug or nutraceutical treatment with potential DMOAD effect (glucosamine, diacerin, chondroitin sulfate) unless given at a stable dose over at least 4 weeks prior to first injection
8. Use of electrotherapy or acupuncture for OA
9. Any known active infections, including suspicion of intra-articular infection and/or infections that may compromise the immune system such as HIV, Hepatitis B or Hepatitis C infection
10. History of sarcoma and/or history of other active malignancy within five years, except adequately treated basal cell and squamous cell carcinoma of the skin
11. Signs and symptoms suggestive of transmissible spongiform encephalopathy
12. Secondary osteoarthritis: e.g. Joint dysplasias, Aseptic osteonecrosis, Acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler's syndrome, Joint infection, Hemophilia, Hemochromatosis, Calcium Pyrophosphate deposition disease, or Neuropathic arthropathy whatever the cause Patients with risk factors for knee OA (e.g. obesity, meniscectomy) are not considered as having secondary OA and can be included in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Nature, incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 24 weeks post treatment
Proportion of subjects with predefined local AEs (acute inflammatory reactions defined as increase of pain by 30 mm - on a 100 mm VAS - associated with a self-reported synovial fluid effusion within 3 days following i.a. injection) | Up to 24 weeks post treatment
Local tolerability in the target knee | Up to 24 weeks post treatment
Laboratory safety parameters (including blood chemistry, haematology, and urinalysis) and ECG | Up to 24 weeks post treatment

SECONDARY OUTCOMES:
Change over time in the levels of the following biomarkers: Biomarkers of anabolic effect on knee cartilage (markers of cartilage formation/synthesis) | Up to 24 weeks post treatment
Change over time in the levels of the following biomarkers: Biomarkers of catabolic effect on knee cartilage (markers of cartilage degradation) | Up to 24 weeks post treatment
Change over time in the levels of the following biomarkers: Biomarkers of Bone Metabolism | Up to 24 weeks post treatment
Change in levels of cytokines related to inflammation (IL1b, IL6, IL8, TNFα and IFNα) | Up to 24 weeks post treatment
Blood levels of AS902330 | Up to 24 weeks post treatment
Presence of anti-AS902330 antibodies | Up to 24 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Donatus Dreher, MD, PhD, Study Director — Merck Serono SA - Geneva
Locations (19):
- UMHAT "Sv. Ivan Rilski", Clinical Research Unit for Phase I, Sofia, Bulgaria
- Denmark (5):
  - Frederiksberg Hospital, Frederiksberg
  - Gentofte Hospital, Hellerup
  - Nordsjællands Hospital - Hørsholm, Hørsholm
  - Silkeborg sygehus, Silkeborg
  - Regionshospitalet Viborg, Viborg
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Turku University Central Hospital, Turku
- South Africa (3):
  - FARMOVS-PAREXEL (Pty) Ltd, University of the Free State, Bloemfontein
  - PAREXEL-George, George
  - PAREXEL-Port Elizabeth, Mercantile Hospital, Port Elizabeth
- Sweden (6):
  - Sahlgrenska University Hospital/Östra, Gothenburg
  - Hässleholms Sjukhus, Hässleholm
  - Kungälv Sjukhus, Kungälv
  - Lund University Hospital, Lund
  - Malmö University Hospital, Malmo
  - Danderyds Sjukhus, Stockholm
- Cambridge University Hospitals, Cambridge, United Kingdom